CLINICAL TRIAL: NCT05928026
Title: Financial Support in an Underserved and Low-Income Population With Heart Failure
Acronym: FUND-HF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Ambarish Pandey, Assistant Professor of Internal Medicine, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STU-2022-1033
Record Dates: First submitted 2023-06-05; First posted 2023-07-03 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Heart Failure, Systolic; Financial Stress; Medication Adherence; Quality of Life
Keywords: social determinants of health
MeSH Terms: conditions — Heart Failure, Systolic; Financial Stress; Medication Adherence | interventions — Financial Support

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate Financial Support (Experimental): This group will receive $500 at the completion of their baseline visit
  Interventions: Behavioral: Financial Support
- Delayed Financial Support (Active Comparator): This group will receive no financial support at their completion of their baseline visit, but will receive $500 at their 1-month visit.
  Interventions: Behavioral: Financial Support

INTERVENTIONS:
Behavioral: Financial Support — A debit card will be loaded with $500 and can be used like a typical debit card.

SUMMARY:
The goal of this clinical trial is to test whether financial support in the form of a one-time $500 stipend would improve medication adherence and quality of life in low-income, socially-needy patients with heart failure with reduced ejection fraction in the post-discharge setting. The main questions it aims to answer are:

* Will financial support improve heart failure quality of life?
* Will financial support improve medication adherence?

Participants will complete surveys on quality of life, social stress, and spending habits at their baseline visit. Participants will be randomly assigned to receive $500 at their baseline visit or $0 at their baseline visit. At their one month visit, quality of life and medication adherence will be assessed. These results will be compared between groups. The group that received $0 at their baseline visit will be provided $500 at their one-month visit and return for a two-month visit. At that visit, quality of life and medication adherence will be assessed. These results will be compared to their one-month results.

Researchers will compare the 1-month quality of life scores and medication adherence scores between the immediate financial support vs delayed financial support. Researchers will also compare 1-month vs 2-month quality of life and adherence data for participants who were randomized to the delayed financial support group.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18
* English speaking participants who completed SOCIAL-HF study surveys
* Ejection Fraction <=40% and eligible for at least one component of GDMT
* Has at least some difficulty paying monthly bills (Somewhat Difficult and Very Difficult)
* Annual household income <130% Federal Poverty Limit
* Have at least two additional social needs based on the following domains:

  * Cost-related nonadherence
  * Food Insecurity
  * Housing Instability
  * Transportation Difficulty
  * Unemployment
  * Household Crowding: Person/Room Ratio >1
  * Rent Burden: Rent/Income Ratio >30%
  * Low social support
  * Interpersonal Violence
  * History of Discrimination

Exclusion Criteria:

* Unwilling to return for 1 and 2-month follow-up visits.
* Currently in jail or prison
* Primary residence outside Dallas County
* Legal Blindness
* Systolic blood pressure <90 mmHg on screening
* Contraindications or Intolerance all medications available for therapeutic drug monitoring (metoprolol, losartan, lisinopril, valsartan, and spironolactone)
* Unable to answer orientation questions.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2023-06-09 (Actual); Primary Completion 2025-04-11 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
Heart Failure Quality of Life by Kansas City Cardiomyopathy Questionnaire (KCCQ) | 1 month
  Quality of life will be ascertained using the KCCQ-12, a validated measure of quality of life among patients with heart failure. The score contains four domains, physical limitation, symptom frequency, quality of life, and social limitations. Each subdomain provides an individual score from 0 to 100, with 0 denoting the worst and 100 denoting the best possible health. These scores are averaged and presented as a summary score.
Heart Failure Quality of Life by Kansas City Cardiomyopathy Questionnaire (KCCQ) | 2 months
  Quality of life will be ascertained using the KCCQ-12, a validated measure of quality of life among patients with heart failure. The score contains four domains, physical limitation, symptom frequency, quality of life, and social limitations. Each subdomain provides an individual score from 0 to 100, with 0 denoting the worst and 100 denoting the best possible health. These scores are averaged and presented as a summary score.

SECONDARY OUTCOMES:
Detection of Serum Levels of Guideline Directed Medical Therapies (GDMT) | 1 month
  This will be ascertained using serum therapeutic drug monitoring of guideline-directed medical therapies.
Self-reported medication adherence by Morisky Medication Adherence Scale | 1 month
  Self-reported medication adherence will be captured by the Morisky Medication Adherence Scale. This scale is an eight-item survey. The score ranges from 0-8, with higher scores denoting greater adherence.
Detection of Serum Levels of Guideline Directed Medical Therapies (GDMT) | 2 months
  This will be ascertained using serum therapeutic drug monitoring of guideline directed medical therapies.
Self-reported medication adherence by Morisky Medication Adherence Scale | 2 months
  Self-reported medication adherence will be captured by the Morisky Medication Adherence Scale. This scale is an eight-item survey. The score ranges from 0-8, with higher scores denoting greater adherence.
Change in social stress | 1 months
  This will be captured using the perceived stress scale. This is a ten-item survey assessing perceived stress over the last month. The scores range from 0-40, with higher scores denoting higher perceived stress.
Change in social stress | 2 months
  This will be captured using the perceived stress scale. This is a ten-item survey assessing perceived stress over the last month. The scores range from 0-40, with higher scores denoting higher perceived stress.

OTHER OUTCOMES:
Psychologic Stress by Kessler Screening Scale | 1 Month
  This is a ten-item instrument measuring psychological distress. Each item has a five-level response scale. The range is 10-50, with higher scores denoting greater psychological distress.
Psychologic Stress by Kessler Screening Scale | 2 months
  This is a ten-item instrument measuring psychological distress. Each item has a five-level response scale. The range is 10-50, with higher scores denoting greater psychological distress.
Number of Emergency Room Visits | 1 Month
  This outcome will be captured through review of the electronic medical record and adjudicated using the DFW Hospital Consortium
Number of Emergency Room Visits | 2 Month
  This outcome will be captured through review of the electronic medical record and adjudicated using the DFW Hospital Consortium
Number of Hospitalizations | 1 Month
  This outcome will be captured through review of the electronic medical record and adjudicated using the DFW Hospital Consortium
Number of Hospitalizations | 2 months
  This outcome will be captured through review of the electronic medical record and adjudicated using the DFW Hospital Consortium
Appointment Completion Rate | 1 Month
  This outcome will be captured through review of the electronic medical records
Appointment Completion Rate | 2 months
  This outcome will be captured through review of the electronic medical records

CONTACTS AND LOCATIONS:
Overall Officials: Ambarish Pandey, MD,MSCS, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Heidenreich PA, Albert NM, Allen LA, Bluemke DA, Butler J, Fonarow GC, Ikonomidis JS, Khavjou O, Konstam MA, Maddox TM, Nichol G, Pham M, Pina IL, Trogdon JG; American Heart Association Advocacy Coordinating Committee; Council on Arteriosclerosis, Thrombosis and Vascular Biology; Council on Cardiovascular Radiology and Intervention; Council on Clinical Cardiology; Council on Epidemiology and Prevention; Stroke Council. Forecasting the impact of heart failure in the United States: a policy statement from the American Heart Association. Circ Heart Fail. 2013 May;6(3):606-19. doi: 10.1161/HHF.0b013e318291329a. Epub 2013 Apr 24. PMID 23616602
- [Background] Greene SJ, Butler J, Albert NM, DeVore AD, Sharma PP, Duffy CI, Hill CL, McCague K, Mi X, Patterson JH, Spertus JA, Thomas L, Williams FB, Hernandez AF, Fonarow GC. Medical Therapy for Heart Failure With Reduced Ejection Fraction: The CHAMP-HF Registry. J Am Coll Cardiol. 2018 Jul 24;72(4):351-366. doi: 10.1016/j.jacc.2018.04.070. PMID 30025570
- [Background] Hood SR, Giazzon AJ, Seamon G, Lane KA, Wang J, Eckert GJ, Tu W, Murray MD. Association Between Medication Adherence and the Outcomes of Heart Failure. Pharmacotherapy. 2018 May;38(5):539-545. doi: 10.1002/phar.2107. Epub 2018 Apr 30. PMID 29600819
- [Background] Wu JR, Moser DK, De Jong MJ, Rayens MK, Chung ML, Riegel B, Lennie TA. Defining an evidence-based cutpoint for medication adherence in heart failure. Am Heart J. 2009 Feb;157(2):285-91. doi: 10.1016/j.ahj.2008.10.001. Epub 2008 Dec 24. PMID 19185635
- [Background] Riegel B, Lee CS, Ratcliffe SJ, De Geest S, Potashnik S, Patey M, Sayers SL, Goldberg LR, Weintraub WS. Predictors of objectively measured medication nonadherence in adults with heart failure. Circ Heart Fail. 2012 Jul 1;5(4):430-6. doi: 10.1161/CIRCHEARTFAILURE.111.965152. Epub 2012 May 30. PMID 22647773
- [Background] Henderson KH, Helmkamp LJ, Steiner JF, Havranek EP, Vupputuri SX, Hanratty R, Blair IV, Maertens JA, Dickinson M, Daugherty SL. Relationship Between Social Vulnerability Indicators and Trial Participant Attrition: Findings From the HYVALUE Trial. Circ Cardiovasc Qual Outcomes. 2022 May;15(5):e007709. doi: 10.1161/CIRCOUTCOMES.120.007709. Epub 2022 Apr 14. PMID 35418247
- [Background] Akwo EA, Kabagambe EK, Harrell FE Jr, Blot WJ, Bachmann JM, Wang TJ, Gupta DK, Lipworth L. Neighborhood Deprivation Predicts Heart Failure Risk in a Low-Income Population of Blacks and Whites in the Southeastern United States. Circ Cardiovasc Qual Outcomes. 2018 Jan;11(1):e004052. doi: 10.1161/CIRCOUTCOMES.117.004052. PMID 29317456
- [Background] Wu JR, Frazier SK, Rayens MK, Lennie TA, Chung ML, Moser DK. Medication adherence, social support, and event-free survival in patients with heart failure. Health Psychol. 2013 Jun;32(6):637-46. doi: 10.1037/a0028527. Epub 2012 Jul 2. PMID 22746258
- [Background] Wu JR, Holmes GM, DeWalt DA, Macabasco-O'Connell A, Bibbins-Domingo K, Ruo B, Baker DW, Schillinger D, Weinberger M, Broucksou KA, Erman B, Jones CD, Cene CW, Pignone M. Low literacy is associated with increased risk of hospitalization and death among individuals with heart failure. J Gen Intern Med. 2013 Sep;28(9):1174-80. doi: 10.1007/s11606-013-2394-4. Epub 2013 Mar 12. PMID 23478997
- [Background] Liao L, Allen LA, Whellan DJ. Economic burden of heart failure in the elderly. Pharmacoeconomics. 2008;26(6):447-62. doi: 10.2165/00019053-200826060-00001. PMID 18489197
- [Background] Barankay I, Reese PP, Putt ME, Russell LB, Loewenstein G, Pagnotti D, Yan J, Zhu J, McGilloway R, Brennan T, Finnerty D, Hoffer K, Chadha S, Volpp KG. Effect of Patient Financial Incentives on Statin Adherence and Lipid Control: A Randomized Clinical Trial. JAMA Netw Open. 2020 Oct 1;3(10):e2019429. doi: 10.1001/jamanetworkopen.2020.19429. PMID 33034639
- [Background] Volpp KG, Loewenstein G, Troxel AB, Doshi J, Price M, Laskin M, Kimmel SE. A test of financial incentives to improve warfarin adherence. BMC Health Serv Res. 2008 Dec 23;8:272. doi: 10.1186/1472-6963-8-272. PMID 19102784
- [Background] Volpp KG, Troxel AB, Mehta SJ, Norton L, Zhu J, Lim R, Wang W, Marcus N, Terwiesch C, Caldarella K, Levin T, Relish M, Negin N, Smith-McLallen A, Snyder R, Spettell CM, Drachman B, Kolansky D, Asch DA. Effect of Electronic Reminders, Financial Incentives, and Social Support on Outcomes After Myocardial Infarction: The HeartStrong Randomized Clinical Trial. JAMA Intern Med. 2017 Aug 1;177(8):1093-1101. doi: 10.1001/jamainternmed.2017.2449. PMID 28654972